CLINICAL TRIAL: NCT07000630
Title: Efficacy and Tolerability of Deucravacitinib in the Management of Palmoplantar Pustulosis; A Nonrandomized Controlled Trial
Brief Title: Efficacy and Tolerability of Deucravacitinib in the Management of Palmoplantar Pustulosis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University First Hospital (Other)
Responsible Party: Principal Investigator, Jingru Sun, Attending doctor, Peking University First Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-452
Record Dates: First submitted 2025-05-24; First posted 2025-06-03 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-05

CONDITIONS: Palmoplantar Pustulosis
Keywords: Palmoplantar pustulosis; Deucravacitinib
MeSH Terms: conditions — Psoriasis | interventions — deucravacitinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Deucravacitinib treatment (Experimental): 25 subjects with palmoplantar pustulosis will be allocated to receive oral Deucravacitinib 6mg everyday for 16 weeks.
  Interventions: Drug: Deucravacitinib

INTERVENTIONS:
Drug: Deucravacitinib — 25 subjects with palmoplantar pustulosis will be allocated to receive oral Deucravacitinib 6mg everyday for 16 weeks.

SUMMARY:
The goal of this clinical trial is to investigate the efficacy and safety of Deucravacitinib in patients with moderate-to-severe palmoplantar pustulosis. Approximately 25 subjects will be included in the study and receive Deucravacitinib 6mg per day for four months. This study will begin June 2025 and is expected to last 14 months.

ELIGIBILITY:
Inclusion Criteria:

* Men and women between ages 18 - 65 years who have suffered from palmoplantar pustulosis (PPP) for at least 6 months.
* Patients were required to have over 10 well-demarcated white or yellow pustules across all regions, with or without plaque psoriasis
* Patients were required to have a Palmoplantar Pustular Physician's Global Assessment (PPPGA) score of at least moderate severity (≥3) and a minimum PPPASI score of 12.
* Signed and dated written informed consent in accordance with ICH GCP and local legislation prior to admission to the trial.
* Further criteria apply.

Exclusion Criteria:

* Systemic treatment for PPP ended less than five half-lives or 12 weeks ago
* Topical treatment for PPP ended less 4 weeks ago
* Women who are pregnant, nursing, or who plan to become pregnant while in the trial.
* Severe, progressive, or uncontrolled condition such as renal, hepatic, haematological, endocrine, pulmonary, cardiac, neurologic, cerebral, or psychiatric disease, or signs and symptoms thereof.
* Presence or known history of anti-TNF-induced PPP-like disease.
* Patient with a transplanted organ (with exception of a corneal transplant >12 weeks Prior to screening) or who have ever received stem cell therapy.
* Known history of lymphoproliferative disease, including lymphoma, or signs and symptoms suggestive of possible lymphoproliferative disease, such as lymphadenopathy and/or splenomegaly.
* Further criteria apply.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2025-06-04 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
Primary efficacy endpoint | From enrollment to the end of treatment at 16 weeks
  The primary efficacy endpoint was percentage change from baseline in Palmoplantar Pustular Area and Severity Index (PPPASI) at W16.

SECONDARY OUTCOMES:
Effect of Deucravacitinib on overall severity of palmoplantar pustulosis | From enrollment to the end of treatment at 16 weeks
  Mean change in erythema and pustules from Baseline to week 16 will be evaluated by Palmoplantar Pustular Physician's Global Assessment (PPPGA).
Effect of Deucravacitinib on quality of life: Dermatology Life Quality Index (DLQI) | From enrollment to the end of treatment at 16 weeks
  Mean change in quality of life from Baseline to week 16 will be evaluated by Dermatology Life Quality Index (DLQI)

OTHER OUTCOMES:
Tolerability of Deucravacitinib in patients with palmoplantar pustulosis | From enrollment to the end of treatment at 16 weeks
  To evaluate the tolerability of Deucravacitinib in patients with palmoplantar pustulosis through assessment of adverse events at every visit from Baseline to week 4, 8,12, 16.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University First Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: Undecided